CLINICAL TRIAL: NCT01908725
Title: A Single-center, Un-controlled, Open-labeled Trial of the Long-term Safety of Lamazym Aftercare Treatment of Subjects With Alpha-Mannosidosis Whom Previously Participated in Lamazym Trials
Brief Title: Lamazym Aftercare Study
Acronym: rhLAMAN-09
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rhLAMAN-09; 2013-000321-31 (EudraCT Number)
Record Dates: First submitted 2013-06-12; First posted 2013-07-26 (Estimated); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Alpha-Mannosidosis
MeSH Terms: conditions — alpha-Mannosidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lamazym (Experimental): 1 mg Lamazym/kg body weight
  Interventions: Drug: Lamazym

INTERVENTIONS:
Drug: Lamazym — ERT, i.v. infusions weekly
  Other Names: rhLAMAN; recombinant human alpha-mannosidase

SUMMARY:
The overall objective of this trial is to provide aftercare treatment with Lamazym and to evaluate the safety of repeated Lamazym i.v. treatment of subjects with alpha-Mannosidosis whom previously participated in Lamazym-trial.

DETAILED DESCRIPTION:
This protocol only concern subjects where compassionate use program was not accepted. Efficacy will be evaluated once yearly to follow the subject's progress in clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* the subject must have participated in previous Lamazym-trials: phase 2b: 2011-004355-40 or phase 3: 2012-000979-17
* Subject or subjects legally authorized guardian(s) must provide signed, informed consent prior to performing any trial-related activities
* The subject and his/her guardian(s) must have the ability to comply with the protocol

Exclusion Criteria:

* Presence of known clinically significant cardiovascular, hepatic, pulmonary, or renal disease or other medical conditions that, in the opinion of the Investigator, would preclude participation in the trial
* Any other medical condition or serious intercurrent illness, or extenuating circumstances that, in the opinion of the Investigator, would preclude participation in the trial
* Pregnancy. Pregnant woman is excluded. Before start fot he treatment the investigators will for women of childbearing potential perform a pregnancy test and decide whether or not there is a need for contraception
* Psychosis; any psychotic disease, also in remission, is an exclusion criteria
* Planned major surgery that, in the opinion of the Investigator, would preclude participation in the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-06; Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Adverse events | 3 year
  AE documented at all visits
Change from baseline in Lamazym antibodies | 3 year
  AB measured every 12th week

SECONDARY OUTCOMES:
progress from baseline in number of steps climbed in 3 minutes | 1 year, 2 year and 3 year
Progress from baseline in equivalent age | 1 year, 2 year and 3 year
Progress from baseline in Forced Vital Capacity | 1 year, 2 year and 3 year
Progress from baseline in distance walked in 6 minutes | 1 year, 2 year and 3 year

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Metabolic Diseases, Department of Clinical Genetics, Juliane Marie Centre, Copenhagen University Hospital, Blegdamsvej 9, Copenhagen, Denmark

REFERENCES:
- See also: 12th international symposium on MPS and related diseases — http://www.google.dk/url?sa=t&rct=j&q=line%20borgwardt&source=web&cd=1&cad=rja&sqi=2&ved=0CCsQtwIwAA&url=http%3A%2F%2Fwww.youtube.com%2Fwatch%3Fv%3DZGgqK7oJQFQ&ei=4TG4UejWD8SSO7TqgbAI&usg=AFQjCNG4azVFYvyGp-yNBeoP4tG6YQQ1Tw&bvm=bv.47810305,d.ZWU
- See also: Results posted in EudraCT — https://www.clinicaltrialsregister.eu/ctr-search/trial/2013-000321-31/results